Title: Communicating multiple disease risks: A translation of risk prediction science

Short title: Comm multi disease risk Aim 2

**Date:** May 4, 2017

**Protocol #: 201706063** 

PI: Erika A. Waters, PhD, MPH 314-747-5705 Washington University School of Medicine Campus Box 8100 660 S. Euclid Ave Saint Louis, MO 63110

Co-I: Ying Liu, Graham Colditz

Consultants: Linda Cameron, Integrity StL, Susan Gillham Design

# **Contents**

| Background and Rationale | 3 |
|----------------------------------|----|
| Objectives | 4 |
| Eligibility Criteria | 4 |
| Registration Procedure | 5 |
| Research Plan | 5 |
| Statistical Considerations | 8 |
| Study Procedure Calendar | 11 |
| Drug Formulation and Procurement | 11 |
| Data and Safety Monitoring Plan | 11 |
| Record Keeping | 12 |
| References | 12 |
| Special Considerations | 15 |
| List of Appendices | 15 |

# **Background and Rationale**

# **RISK CALCULATOR (Parent grant)**

Epidemiology seeks to improve public health by identifying risk factors for cancer and other diseases and conveying that information to relevant audiences (e.g., physicians, the public). The audience is presumed to understand and use that information to make appropriate decisions about lifestyle behaviors and medical treatments. Yet, even though a single risk factor can affect the risk of multiple health outcomes, this information is seldom communicated to people in a way that optimizes their understanding of the importance of engaging in a single healthy behavior. [1] Providing individuals with the ability to understand how a single behavior (obtaining sufficient physical activity) could affect their risk of developing multiple diseases could foster a more coherent and meaningful picture of the behavior's importance in reducing health risks, and increase motivation and intentions to engage in the behavior.

We will test the effectiveness of a risk calculator that conveys individualized risk estimates for colon cancer, heart disease, diabetes, stroke, and breast cancer (women) to socio-demographically diverse laypeople who do not get 150 minutes of moderate intensity physical activity per day. Estimates of how the participant's risk would change if they were to engage in at least 3 hours of moderate intensity activity per week will also be provided.

# **MENTAL IMAGERY (Supplement)**

Although risk calculators can improve comprehension and produce favorable changes in health cognitions that lead to behavior change (e.g., accuracy of perceived risk, response efficacy, intentions), the effect of calculators on behavior itself is modest. [2-4] However, the gap between intentions and behavior can be bridged via interventions that help people develop self-regulatory skills, such as developing action plans for how to achieve each step of the behavior. [5-8] Mental imagery may be particularly useful in the development and realization of these plans. [5, 9, 10]

We will adapt an existing and effective mental imagery-based self-regulation physical activity intervention<sup>[5]</sup> for incorporation into the working risk calculator and compare its effectiveness in increasing physical activity behavior to an active control that addresses sleep hygiene.

# RISK CALCULATOR AND MENTAL IMAGERY (Conceptual Model)

The conceptual model was adapted from the Health Action Process Approach (HAPA).[8] It asserts that behavior change occurs in two phases. The motivation phase is most relevant for people who do not engage in the recommended behavior. The goal of interventions that target the motivation phase – such as the risk calculator – is to increase intentions to engage in the behavior. Risk perceptions are important in this phase because they raise awareness of the consequences of not engaging in the behavior. Together with outcome expectancies (e.g., the expected consequences of engaging in the behavior, operationalized here as response efficacy), perceived severity of the health outcome, and action self-efficacy (i.e., confidence in one's ability to initiate a new behavior), risk perceptions influence intentions to start the behavior change process. Note that the risk calculator is not expected to increase action self-efficacy or perceived severity because it was not designed with a component to target those constructs.

We enhanced the motivation phase of the conceptual model with additional components drawn from risk perception and communication research. Comprehension of information was added because perceptions and comprehension are slightly different constructs that each have an important role in influencing health behavior and decisions.[11] Worry, affective reaction to the information, affective attitudes to exercise, and anticipated regret were added because a growing body of research demonstrates that affect and emotion are integral to the formation of risk perceptions, in increasing motivation to change behavior, and in changing behavior itself.[12-17] Demographics, numeracy, health literacy, and graph literacy were added because they are associated with the ability to understand and use health risk information. [18-20]

According to HAPA, progression to the action phase is dependent upon factors not included in the motivation phase. These new factors include developing action plans for engaging in the behavior, coping plans for overcoming barriers to action, maintenance self-efficacy (i.e., confidence in the ability to overcome barriers to acting), and recovery self-efficacy (i.e., confidence in the ability to recover from a relapse).

# **Objectives**

#### **RISK CALCULATOR**

To compare the effectiveness of communicating personalized risk estimates via text, table, or risk ladder.

Primary outcomes hypotheses and exploratory research questions

- H1: Comprehension of risk information and intentions to increase physical activity will be higher among individuals who see multiple disease risks presented as a risk ladder than as text.
- RQ1: Prior research has shown that tables can be effective in communicating risk information. [21] Compared to the table, will the risk ladder elicit higher comprehension and intentions?

Secondary outcomes hypotheses and exploratory research questions

- H2: Any significant effect of the risk ladder on intentions will be mediated by comprehension, risk perceptions, response efficacy, worry, affective reactions to information, affective attitudes to exercise, and anticipated regret.
- H3: Engagement in physical activity will increase from baseline to 90 day follow-up to a greater extent for individuals who see the risk ladder than those who see text only.
- H4: Intentions will mediate any significant effect of the risk ladder on physical activity.
- RQ2: Compared to the table, will the risk ladder elicit higher risk perceptions, response efficacy, worry, affective reactions to information, affective attitudes to exercise, and anticipated regret?

Sociodemographic exploratory research questions

RQ3: Will education, race/ethnicity, numeracy, health literacy, and/or graph literacy moderate the effect of risk communication strategy on primary outcomes?

#### MENTAL IMAGERY

To test whether supplementing the risk calculator with a mental imagery-based self-regulation intervention will increase actual engagement in physical activity over time, and to explore several possible mechanisms.

Primary outcome and exploratory research questions

- H5: Engagement in physical activity will increase from baseline to 90-day follow-up only among individuals in the physical activity mental imagery intervention, [5, 7-9] not in the sleep hygiene imagery active control condition.
- RQ5: Will education, race/ethnicity, numeracy, health literacy, and/or graph literacy moderate the effect of mental imagery condition on behavior?

Secondary outcomes and exploratory research questions

- H6: Within the physical activity mental imagery condition, increases in activity from pre-intervention baseline to 90-day follow-up will be preceded by the following measures assessed at the week 4 follow-up: action planning, coping planning, action self-efficacy, maintenance self-efficacy, recovery self-efficacy, affective attitudes to exercise, and perceived vividness of imagery. [5, 7-9, 16]
- RQ6: Within the physical activity mental imagery condition, the direction and magnitude of change in activity from pre-intervention baseline to week 1 follow-up will be preceded by the following measures assessed at the survey assessed immediately post-intervention: action planning, coping planning, action self-efficacy, maintenance self-efficacy, recovery self-efficacy, affective attitudes to exercise, and perceived vividness of imagery. [5, 7-9, 16] Similarly, measures assessed at week 1 will predict change in behavior from week 1 to week 2; measures assessed at week 2 will predict behavior change from week 2 to week 3: and measures assessed at week 3 will predict behavior change from week 3 to week 4.

# **Eligibility Criteria**

#### RISK CALCULATOR AND MENTAL IMAGERY

Inclusion criteria are: 30-64 years of age, less than three relevant comorbidities (diabetes, heart disease, stroke and cancer, where cancer counts as 2 comorbidities for women but 1 for men due to the statistical properties of the risk calculator), having a SMS/text capable mobile phone that is not shared with anyone else, text messaging more than once a month, and not meeting national guidelines for aerobic physical activity (i.e., at least 150 minutes per week of moderate intensity aerobic physical activity).[22]

# **Registration Procedure**

#### RISK CALCULATOR AND MENTAL IMAGERY

Participants will be recruited from the Recruitment Enhancement Core (REC), reasearchmatch.org, the Health Communication Research Lab's FReDa database, word of mouth, newspaper advertisements, and a database maintained by the Waters Lab. REC will follow their established standard procedures by posting information about the study in BJC today (Appendix P: Aim 2, BJC Ad), on the REC website (Appendix T: Aim 2, Website posting), Facebook (Appendix R: Aim 2, Facebook Posting), Centerwatch (Appendix Q: Aim 2, Centerwatch Ad), and newspaper advertisements (Appendix CC, Newspaper Advertisement). REC will forward interested participants' contact information to the study team, who will make outbound calls to potential participants. Researchmatch.org will email registry members with information about the study (Appendix U: Aim 2, Researchmatch.org email), and offer participants a chance to contact the study team if they are interested in participating. The study team will make outbound calls and emails to members of the HCRL FReDa database and Waters Lab database (Appendix N: Aim 2, Screening Call Script; Appendix O: Aim 2, Recruitment Email Script).

In addition, we will also recruit participants in person at various locations around St. Louis. The locations will be determined by the REC and will include publicly available places with private space available, like laundromats, libraries, and community centers. In this case, research assistants will speak with potential participants in person to assess interest in the study. If potential participants are interested in participating in the study, research assistants will go through appendix H, the eligibility screener. If the participant is eligible, the study team member will record the participant's contact information on Appendix I, the Contact Info Sheet. If the participant is able to conduct the data collection session immediately, the research assistant will continue on to begin the data collection session following Appendix W (Aim 2 Data collection session 1 guide). If the participant is not able to conduct the data collection session immediately, we will schedule a time for the session at a later date, or offer times for walk-in sessions. Study coordinators will schedule sessions to take place either at the Taylor Avenue Building (Wash U) or at a mutually agreed upon public place with adequate private space to conduct the interview (e.g. a meeting room at a library). When the participant arrives for the session, the research assistant will explain the study procedures, obtain written consent, and begin data collection.

We will enroll 500 participants. Recruitment will be stratified based on race (at least 50% racial/ethnic minority) and education (at least 50% will have no college experience) to ensure adequate representation of populations that experience health disparities and, consequently, to increase relevance of the intervention to those groups.

#### Research Plan

## **RISK CALCULATOR AND MENTAL IMAGERY**

## Design

This study will use a 3 (risk presentation condition: text vs. table vs. risk ladder) x 2 (mental imagery condition: physical activity vs. sleep hygiene) experimental design. Participants will be block randomized to ensure that each of the 6 experimental conditions has equal numbers of participants at the end of the study. Randomization will occur by the computer program after eligibility screening and consent, but prior to engaging in any study activities.

Blinding

The research staff will be blinded to participants' risk presentation conditions, but they will unblinded to mental imagery condition. This unblinding was the result of a combination of the block randomization (which prevented us from preparing packets of study materials ahead of time and assigning participants to condition in order of completion (e.g., A, B, C, D, E, F)), and the need for the goal cards and Baseline Survey 2 to include information specific to the mental imagery condition the participant was assigned to (see below).

#### Procedure

The procedures for the study will occur in 3 parts. Part 1 is an initial 45 minute data collection session in person, followed by (Part 2) reminders and surveys conducted by Short Message Service (SMS) text messaging over the subsequent 4 weeks, and (Part 3) a final mailed survey on paper. The last half of Part 1 and all of Part 2 are adapted from prior research conducted by Linda Cameron for use with University of Auckland employees. [5, 9] We worked closely with Dr. Cameron to adapt the interventions so they would be acceptable to our St. Louis community sample (e.g., minimize burden, reduce the need for Internet access, to accommodate cell phone plans that do not have unlimited text and/or data, etc). This adaptation was performed in Spring 2017 and involved 3 sets of cognitive interviews, each set including 6-7 participants (Aim 2, Part 1).

Part 1, Baseline Intervention Administration and Data Collection. Participants will complete all baseline activities in person with a research assistant. After completing eligibility screening and informed consent processes, participants will use a smartphone provided by research staff to complete the risk calculator portion of the study. The research assistant will enter the participant ID into the responsive website, and then the participant will provide information about their demographics, health behaviors, and personal and family health history (Appendix A Aim 2, Risk Display App Screens, pg. 2-34). The website then provides participants with personalized risk results for their current activity level and how it would change if they began exercising regularly. Results are displayed either as alphanumeric text, table, or risk ladder (Appendix A Aim 2, Risk Display App Screens, pg. 35-38). Afterwards, the participant will complete Baseline Survey 1 independently on paper (Appendix C, Instructions Appendix HH).

Immediately after completing Baseline Survey 1, participants will begin the mental imagery component of the study. The research assistant will enter the participant's personal phone number into the website so they can receive text messages for the next 4 weeks. Then, participants will use the smartphone and headphones provided by the research team to listen to an audiorecording that walks the participant through how to set a physical activity or sleep goal and asks them to imagine themselves exercising or improving their sleep hygiene (Appendix A Aim 2, Risk Display App Screens, pg. 39-42; Appendices D and E, Mental Imagery audio recording scripts). Participants will be asked to practice this mental imagery twice a day for 5 minutes each day the subsequent weeks. The audio recording also instructs the participant to write down an exercise or sleep-related goal on a pamphlet provided by the research assistant (Appendix F, Pamphlet). Participants will then complete Baseline Survey 2 independently on paper (Appendices L and M). Based on the cognitive interviews conducted in Spring, 2017, Part 1 will take approximately 45 minutes. Participants will receive a \$20 gift card to Schnucks for their time and effort.

Part 2. SMS/Text Message Intervention and Data Collection. Beginning at 7:00pm on the day the participant completes the Baseline/Part 1 activities, the participant will begin receiving text messages related to the study. The first texts will welcome them to the study and provide information about how to contact the Lab, how to stop the texts from being sent, and how to access the audiorecording to which they were assigned (physical activity vs. sleep). At noon on Mondays, Wednesdays, and Fridays, they will be sent 1 of 3 texts that remind them to practice the imagery presented in the audio recording twice daily for five minutes each time. These reminders will continue for 3 weeks. Each week after the 3<sup>rd</sup> reminder they will receive a text message based survey. A final text message based survey will be sent one week after the third text message based survey. The content and schedule for the text messages and text surveys are found in Appendices X and Y (Text Message Reminders and Survey- Exercise, Sleep). Each text message length is no more than 160 characters, including spaces, to fit within the universal constraints of SMS messaging protocols. This was done to avoid having 1 intended message being sent in multiple pieces. The total participation time per week is estimated to be approximately 10 minutes. Participants will earn a \$10 gift card to Schnucks for each text message survey they complete. This amount is intended to help offset the cost of text messages for participants who may not have unlimited text messaging.

Part 3, Mailed 90-Day Follow-Up Survey. Ninety days after Baseline/Part 1, participants will receive a final follow-up study survey (Appendix BB) in the mail along with a written survey invitation (Appendix AA). If participants do not complete the first mailed survey, we will follow-up with one reminder call (Appendix Z) and one additional mailed survey. The survey is expected to take approximate 15 minutes. Participants will receive a \$20 gift card for Schnucks for completing the follow-up survey.

Part 4, Follow-Up Phone Call. Within one year of the final follow up period, we may contact up to 20 participants by phone and ask them questions about their experience and thoughts on the study process (Appendix II). If this occurs, the phone call will take approximately 10 to 15 minutes.

#### Measures

Baseline Survey 1

(Appendix C)

To reduce participant burden, we limit the number of survey questions by adapting single item measures used in nationally representative surveys and in published empirical research. Many items are identical or very similar to the items in Aim 1 and Aim 2, Part 1 of the study. All items for the proposed research, including items that were adapted or developed specifically for Aim 2, Part 2, underwent cognitive testing in either Aim 2, Part 1 or in prior research studies conducted by the Waters Lab. Adaptations to the items intended for use in the text messaging surveys (160-character limit) were made in close collaboration with Linda Cameron, who was the initial developer of the interventions. Table 1 below provides each of the measures that will be assessed in each part of the survey.

Questionnaire Name Timing Content Part 1: Baseline Eligibility Screener Pre-randomization Age; [23] race/ethnicity; [23] education; [23] personal diagnosis of the target diseases; [24, 25] physical activity behavior; [26, 27] and cell phone (Appendix H) access (developed in-house) Risk Assessment Immediately following Demographic, biological, and behavioral characteristics needed for the risk algorithm<sup>[28-30]</sup> (Appendix A) randomization to 1 of

6 conditions in a 3 (risk presentation: text vs. table vs. risk ladder) x 2 (mental imagery: physical activity vs. sleep hygiene) design

Table 1. Summary of Study Measures, in Order of Completion

Immediately following provision of personalized risk information

Comprehension:<sup>[31]</sup> cognitive and affective perceived risk;<sup>[32]</sup> perceived severity[33] worry;[32] response efficacy;[34] action selfefficacy;[35] affective reaction to the information;[36] affective attitude about exercise;[16] anticipated regret;[17] intentions to engage in physical activity in the next 90 days;[34] numeracy[37]; graph literacy;[20] health literacy.[38] self-reported health status;[24] work schedule;[39] sleep behavior. [9] Other items intended to be used as preliminary data in future studies examining possible defensive processing of personalized health risk information include: perceived accuracy of information; [4, 40] message acceptance; [41] defensive processing [42] time orientation,<sup>[43]</sup> and spontaneous self-affirmation.<sup>[32]</sup>

# Baseline Survey 2 (Appendices L and M)

Immediately following completion of the mental imagery activity. The specific item wording is tailored based on which mental imagery condition is assigned (i.e., mental imagery vs. sleep), but the constructs assessed are the same for both conditions.

Message acceptance,<sup>[41]</sup> perceived clarity and vividness of images;<sup>[5, 9]</sup> and the following items obtained, developed, or adapted from:<sup>[5, 6, 9, 34]</sup> action plan; coping plan; action self-efficacy; recovery self-efficacy; and maintenance self-efficacy.

# Part 2: Text Messaging

Mid-Intervention Text Message Surveys (Appendices X and Y) 1, 2, 3, and 4 weeks after Part 1

Perceived clarity and vividness of images; [5, 9] and the following items obtained, developed, or adapted from: [5, 6, 9, 34] action plan; coping plan; action self-efficacy; recovery self-efficacy; and maintenance self-efficacy.

# Part 3: 90-Day Follow-Up

Follow-Up (Appendix BB)

90 days after Part 1

Comprehension;<sup>[31]</sup> physical activity behavior,<sup>[26, 27]</sup> sleep behavior,<sup>[9]</sup> tobacco use,<sup>[27]</sup> and the same items as in Baseline Survey 2 assessing intentions, action self-efficacy, cognitive and affective perceived risk, response efficacy, anticipated regret, and affective attitudes.

<u>Note:</u> Race and education will be assessed during eligibility for recruitment stratification purposes only. Baseline Survey 1 excludes characteristics that will be assessed in the Risk Assessment questionnaire.

#### **Statistical Considerations**

#### Preliminary Analyses

We will begin by using descriptive statistics to understand the frequency and distributional properties of all items. For variables with non-normal distributions, data transformations or non-parametric tests will be used for subsequent analyses.

Cronbach  $\alpha$  will be used to test the internal consistency of multi-item constructs in Baseline Survey 1 (i.e., cognitive and affective perceived risk; response efficacy; action self-efficacy; affective reaction to the information; affective attitude about exercise; anticipated regret; intentions to engage in physical activity, message acceptance), Baseline Survey 2 (i.e., message acceptance, perceived clarity and vividness of images), and the Follow-Up Survey (i.e., intentions, action self-efficacy, cognitive and affective perceived risk, response efficacy, anticipated regret, affective attitude about exercise). Where  $\alpha \ge .70$  we will create a scale by averaging responses to a given construct across diseases. That average score will be used in subsequent analyses. Comprehension, numeracy, and graph literacy will each be operationalized as continuous variables comprised of the number of items answered correctly.

Next, we will verify that participant characteristics (i.e., demographics, personal diagnosis of one of the target Communicating Multiple Disease Risk, Aim 2, Part 2 (Version 1) 8

diseases, self-reported health status, numeracy, health literacy, graph literacy, pre-intervention minutes of physical activity per week) are equivalent across experimental conditions by conducting t-tests, one-way ANOVAs, chi-square tests, or other tests, as appropriate. If any differences are found, these variables will be included in subsequent analyses as potential covariates. Personal characteristics will also be explored to determine if they are related to the outcomes of interest. Any characteristic that has a significant association with the outcomes will be included in subsequent analyses as potential covariates.

## Main Analyses

All hypotheses and research questions will be examined using separate analyses for each outcome variable. Assumptions of each type of test will be checked (e.g., assumptions of normality and homogeneity of variance for ANOVAs). If there are violations, non-parametric tests will be used instead. Sex will be a covariate because there are no valid prediction models for male breast cancer, so men will not be shown a breast cancer risk estimate. The inclusion of other personal characteristics as covariates will be determined by the results of the preliminary analyses. Tests of moderation will be conducted by creating interaction terms between the risk presentation condition or mental imagery condition variables, as appropriate, and the variable assessing the moderator of interest. All statistical tests will be based on list-wise deletion except structural equation models, which can accommodate missing data.

Mediation analyses will be conducted using structural equation modeling (SEM). Full Information Maximum Likelihood estimation (FIML)[44] will be used to allow the inclusion of missing data. Standardized estimates will be calculated and bias-corrected bootstrapping will be used to obtain the 95% confidence intervals. [45-48] Criteria assessing model fit will also be examined (e.g., Standardized Root Mean Square Residual ≤.08, comparative fit index ≥.95, root mean square error of approximation ≤.06). [49, 50] Mediational analyses will examine each construct as an individual mediator first, and then as a multiple mediator model.

Table 2 below describes the analyses that will be conducted for each hypothesis or research question.

| Table 2. Overview of Statistical Analyses | | | | |
|---|---|---|---|---|
| | Priority | Statistical test(s) | Outcomes | Predictors/Mediators/Moderators |
| Risk | Calculator | | | |
| H1;<br>RQ1 | Primary | 3 arm ANOVA, 2<br>planned contrasts<br>(risk ladder vs. text;<br>risk ladder vs.<br>table) | Comprehension, intentions | Predictor: Risk presentation condition |
| H2 | Secondary | condary SEM Intentions | | <u>Predictor:</u> Risk presentation condition (risk ladder vs. text) |
| | | | | Mediators: comprehension, risk perceptions, response efficacy, worr affective reactions to information, affective attitudes to exercise, anticipated regret |
| НЗ | Secondary | 3 arm ANOVA,<br>planned contrast<br>(risk ladder vs. text) | Change in physical activity<br>(mins/week at 90 days –<br>mins/week at baseline) | Predictor: Risk presentation condition |
| H4 | Secondary | SEM | Change in physical activity (mins/week at 90 days – mins/week at baseline) | <u>Predictor:</u> Risk presentation condition (risk ladder vs. text) <u>Mediator:</u> Intentions |
| RQ2 | Secondary | 3 arm ANOVA,<br>planned contrast<br>(risk ladder vs. | Risk perceptions, response efficacy, worry, affective reactions to information, affective attitudes | Predictor: Risk presentation condition |

| | | , | , , | |
|---|---|---|---|---|
| RQ3 | Secondary | 3 arm ANOVA | Comprehension, intentions | Predictor: Risk presentation condition Moderators: Education, race/ethnicity, numeracy, health and graph literacy |
| Menta | al Imagery | | | |
| H5 | Primary | T-test | Change in physical activity<br>(mins/week at 90 days –<br>mins/week at baseline) | <u>Predictor:</u> Mental imagery condition |
| RQ5 | Primary | ANOVA | Change in physical activity<br>(mins/week at 90 days –<br>mins/week at baseline) | <u>Predictor:</u> Mental imagery condition<br><u>Moderators:</u> Education, race/ethnicity,<br>numeracy, health and graph literacy |
| H6 | Secondary | Regression<br>(physical activity<br>mental imagery<br>condition only) | Change in physical activity<br>(mins/week at 90 days –<br>mins/week at baseline) | Predictors: Week 4 action planning, coping planning, action self-efficacy, maintenance self-efficacy, recovery self-efficacy, affective attitudes to exercise, perceived vividness |
| RQ6 | Secondary | Regression<br>(physical activity<br>mental imagery<br>condition only) | Weekly change in minutes of<br>physical activity, assessed by 4<br>difference scores: Week1-<br>Baseline; Week2-Week1; Week3-<br>Week2; and Week4-Week3 | Predictors: For each weekly behavioral assessment, use the previous week's measures of the following constructs: action planning, coping planning, action self-efficacy, maintenance self-efficacy, recovery self-efficacy, affective attitudes to exercise, perceived vividness. |

to exercise, anticipated regret

#### Sample Size Calculations

table)

We will enroll 500 participants at baseline. This will enable us to test the primary hypothesis for each of the components of the study. This calculation was based on the information below.

#### **RISK CALCULATOR**

Sample size was calculated to be able to detect an effect of risk presentation strategy on the primary outcome variables comprehension and intentions (Risk Calculator Hypothesis 1 and RQ1). Based on a 2-sided test of means for 3 groups (ANOVA) at 80% power,  $\alpha$ =.05, df=2, and Cohen's f effect size of 0.15 (approximately equivalent to Cohen's d of 0.3),<sup>[51, 52]</sup> we anticipate needing 432 participants. The effect size estimate was based on a study of personalized breast cancer risk and risk reduction communication that found an effect on intentions to increase physical activity of approximately f=0.25 and an effect on response efficacy of approximately f=0.20.<sup>[4]</sup> However, most of those participants were white, highly educated, had high health literacy, and recruited from a breast health center. Thus, we can expect the findings in our more diverse sample to be somewhat lower. We chose f=.15 as a reasonable compromise because it represents slightly more than a minimal effect,<sup>[53]</sup> but is also logistically feasible. To account for the possibility of 10% missing data in Baseline Survey 1, which assesses the constructs for the Risk Calculator Hypothesis 1, we would need to enroll 480 participants to obtain 432 completed surveys.

#### **MENTAL IMAGERY**

Dr. Cameron's prior self-regulatory intervention accounted for approximately 20% of the unique variance in physical activity at 4-week follow-up. This is approximately equivalent to a Cohen's d effect size of 1.0, which is considered a large effect. Because our follow-up is 90 days, we can expect that our effect size will be somewhat lower. Other self-regulation interventions yielded smaller effects over varying timeframes (e.g., d=0.28-0.78). Thus, powering the study to detect an effect of d=0.30 of the intervention on behavior (Mental

Imagery Hypothesis 5) would be conservative and reasonable. Based on a 2-sided test of means for 2 groups (t-test) at 80% power,  $\alpha$ =.05, and Cohen's d effect size of 0.30, $^{[51,52]}$  we anticipate needing 352 participants at 90-day follow-up. To account for the possibility of 30% attrition rate due to our underserved sample (unpublished data), we expect needing to enroll 500 participants at baseline to achieve this goal.

# **Study Procedure Calendar**

| Table 3. Study Timeline | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Year 1 | | | | Year 2 | | | Year 3 | | | | Year 4 | | | | |
| | 1 | 2 | 3 | 4 | 1 | 2 | 3 | 4 | 1 | 2 | 3 | 4 | 1 | 2 | 3 | 4 |
| Startup (hiring, IRB amendments) | Χ | Χ | Χ | Χ | | | | | Χ | | | | | | | |
| Biweekly research team meetings | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ |
| Aim 1, Part 1: modify and refine stimulus (includes cognitive interviews) | Х | Х | Х | | | | | | | | | | | | | |
| Aim 1, Part 2: refine, program, pilot test, and finalize questionnaires | Х | Х | Х | | | | | | | | | | | | | |
| Aim 1, Part 2: collect data (GfK) | | | | Χ | | | | | | | | | | | | |
| Aim 1, Part 2: analyze and interpret data | | | | | Χ | Χ | Х | | | | | | | | | |
| Aim 1, Part 2: disseminate results | | | | | | | Х | Χ | Χ | Χ | | | | | | |
| Aim 2, Part 1: convert relative risk | Х | Х | Χ | Χ | | | | | | | | | | | | |
| estimates to absolute risk estimates | | | | | | | | | | | | | | | | |
| Aim 2, Part 1: disseminate results | | | | Х | X | X | | | | | | | | | | |
| Aim 2, Part 1: write and verify the accuracy of the computer code used to | | | | | Х | X | X | X | | | | | | | | |
| calculate risk estimates and show the risk results displays (includes interviews) | | | | | | | | | | | | | | | | |
| Aim 2, Part 2: Recruit participants and | | | | | | | | | Χ | Χ | Х | Х | | | | |
| implement risk calculator and mental | | | | | | | | | | | | | | | | |
| imagery interventions | | | | | | | | | | | | | | | | |
| Aim 2, Part 2: 90-day follow-up | | | | | | | | | | Х | Х | Χ | Х | | | |
| Aim 2, Part 2: analyze data | | | | | | | | | | | | Х | Χ | Χ | | |
| Aim 2, Part 2: disseminate results | | | | | | | | | | | | | | | Χ | Χ |

# **Drug Formulation and Procurement**

Not applicable.

#### **Data and Safety Monitoring Plan**

## **RISK CALCULATOR AND MENTAL IMAGERY**

#### Voluntary participation

We will protect against emotional discomfort by emphasizing that participation is voluntary. Participants will provide informed consent. They will be informed that participation is voluntary and that they can elect not to answer any question that makes them uncomfortable or withdraw at any time during the study without any penalty. Additionally, participants will be informed that all study data will be kept confidential and that all personal identifiers will be destroyed when the study is completed.

## Confidentiality and Data Security

There are several layers of protection regarding confidentiality and data security.

First, the study is undergoing a Washington University Information Security Office IRB Study Security review. A detailed description of our study's confidentiality and data security features is described in that document. (see Appendix JJ).

Second, the websites that host the data (i.e., Amazon Web Services and Twilio) have extensive security precautions. These precautions are being reviewed by the Information Security Office (see Appendices JJ, KK, and LL).

Third, the study team will be alert for any potential breaches to prevent inadvertent release of confidential information. If a potential breach in confidentiality occurs, the PI will work with the Institutional Review Board, HIPAA, and the Information Security Office according to their rules and regulations for such a situation.

Fourth, all study data will be downloaded to WUSM servers on a daily basis. Access to data will be password protected to restrict use by non-study personnel. All data will be stored using ID numbers, not names. Participants' responses to study questions will be coded to protect their confidentiality, and names will be kept separate from survey data. Any data that is transported on portable storage devices will be encrypted. Hard copies collected at the in person recruitment locations will be transferred to storage by an RA in a closed envelope and will not leave sight of the RA until securely stored. All paper copies will be will be stored in a locked filing cabinet in a locked suite in an entry controlled building. No personally identifying information will appear in any presentations or publications that results from this study; only aggregated data will be disseminated.

# **Record Keeping**

#### RISK CALCULATOR AND MENTAL IMAGERY

Records will be maintained by the study coordinator and supervised by the PI. All information will be recorded in password-protected databases and held on WUSM servers, which are encrypted and backed up nightly. The study coordinator will record the following pieces of information:

- Participants' contact information, which is needed for the text messaging and follow up activities (i.e., Parts 2 and 3).
- Survey responses, which are linked to participants via an individual identifier but are not linked to names or contact information.

Paper copies of study materials will be kept in a locked filing cabinet located within a locked office suite. For additional information, see <u>Data Safety and Monitoring Plan</u>.

#### References

- 1. Waters EA, Sullivan HW, Nelson W, Hesse BW. What is my cancer risk? Identifying how Internet-based cancer risk calculators convey individualized risk estimates to the public. J Med Internet Res. 2009;11(3):e33. doi: http://dx.doi.org/10.2196/jmir.1222. PMCID: PMC2762854.
- 2. Sheeran P, Harris PR, Epton T. Does Heightening Risk Appraisals Change People's Intentions and Behavior? A Meta-Analysis of Experimental Studies. Psychol Bull. 2013. doi: 10.1037/a0033065.
- 3. Webb TL, Sheeran P. Does changing behavioral intentions engender behavior change? A metaanalysis of the experimental evidence. Psychol Bull. 2006;132(2):249-68.
- 4. Fowler SL, Klein WM, Ball L, McGuire J, Colditz GA, Waters EA. Using an Internet-Based Breast Cancer Risk Assessment Tool to Improve Social-Cognitive Precursors of Physical Activity. Med Decis Making. 2017:272989X17699835. doi: 10.1177/0272989X17699835.
- 5. Chan CK, Cameron LD. Promoting physical activity with goal-oriented mental imagery: a randomized controlled trial. J Behav Med. 2012;35(3):347-63. doi: 10.1007/s10865-011-9360-6.
- 6. Gollwitzer PM. Implementation intentions: Strong effects of simple plans. Am Psychol. 1999;54(7):493-503.
- 7. Gollwitzer PM, Sheeran P. Implementation intentions and goal achievement: A meta-analysis of effects and processes. Adv Exp Soc Psychol. 2006;38:69-119.
- 8. Schwarzer R. Social-cognitive factors in changing health-related behavior. Curr Dir Psychol Sci. 2001;10(2):47-51.
- 9. Loft MH, Cameron LD. Using mental imagery to deliver self-regulation techniques to improve sleep behaviors. Ann Behav Med. 2013;46(3):260-72. doi: 10.1007/s12160-013-9503-9.

- 10. Martin KA, Moritz SE, Hall CR. Imagery use in sport: A literature review and applied model. The Sport Psychologist. 1999;13:245-68.
- 11. Weinstein ND. What does it mean to understand a risk? Evaluating risk comprehension. J Natl Cancer Inst Monogr. 1999;25(1):15-20.
- 12. Finucane ML, Alhakami A, Slovic P, Johnson SM. The affect heuristic in judgments of risks and benefits. J Behav Decis Mak. 2000;13(1):1-17.
- 13. Janssen E, Waters EA, van Osch L, Lechner L, de Vries H. The importance of affectively-laden beliefs about health risks: the case of tobacco use and sun protection. J Behav Med. 2012. Epub 2012/10/18. doi: 10.1007/s10865-012-9462-9. PMCID: PMC4101804.
- 14. Hay J, McCaul KD, Mangan RE. Does worry about breast cancer predict screening behaviors? A metaanalysis of the prospective evidence. Preventive Medicine: An International Journal Devoted to Practice and Theory. 2006;42(6):401-8.
- 15. Kiviniemi MT, Rothman AJ. What do people think about changes in health behaviors? Differential perceptions of consequences of increases and decreases in health behaviors. Psychol Health. 2008;23(7):867-85. Epub 2009/10/06. doi: 10.1080/14768320701360500. PMCID: PMC2753289.
- 16. Kiviniemi MT, Voss-Humke AM, Seifert AL. How Do I Feel About the Behavior? The Interplay of Affective Associations With Behaviors and Cognitive Beliefs as Influences on Physical Activity Behavior. Health Psychol. 2007;26(2):152-8.
- 17. Weinstein ND, Kwitel A, McCaul KD, Magnan RE, Gerrard M, Gibbons FX. Risk perceptions: Assessment and relationship to influenza vaccination. Health Psychol. 2007;26(2):146-51.
- 18. Nelson W, Reyna VF, Fagerlin A, Lipkus I, Peters E. Clinical implications of numeracy: Theory and practice. Ann Behav Med. 2008;35:261-74.
- 19. Nelson WL, Moser RP, Han PK. Exploring objective and subjective numeracy at a population level: findings from the 2007 Health Information National Trends Survey (HINTS). Journal of health communication. 2013;18(2):192-205. doi: 10.1080/10810730.2012.688450.
- 20. Galesic M, Garcia-Retamero R. Graph Literacy: A Cross-Cultural Comparison. Med Decis Making. 2011;31(3):444-57. Epub 2010/07/31. doi: 0272989X10373805
- 21. Schwartz LM, Woloshin S. The Drug Facts Box: Improving the communication of prescription drug information. Proc Natl Acad Sci U S A. 2013;110 Suppl 3:14069-74. doi: 10.1073/pnas.1214646110. PMCID: PMC3752172.
- 22. Garber CE, Blissmer B, Deschenes MR, Franklin BA, Lamonte MJ, Lee IM, Nieman DC, Swain DP, American College of Sports M. American College of Sports Medicine position stand. Quantity and quality of exercise for developing and maintaining cardiorespiratory, musculoskeletal, and neuromotor fitness in apparently healthy adults: guidance for prescribing exercise. Med Sci Sports Exerc. 2011;43(7):1334-59. doi: 10.1249/MSS.0b013e318213fefb.
- 23. Knowledge Networks. Core Adult Profile Survey. 2012.
- 24. National Cancer Institute. Health Information National Trends Survey (HINTS) items for years 2003-2007 Bethesda, MD: National Cancer Institute; 2009 [cited 2010 June 7]. Available from: <a href="http://hints.cancer.gov/questions/all-guestions1.jsp">http://hints.cancer.gov/questions/all-guestions1.jsp</a>.
- 25. National Center for Health Statistics. National Health Interview Survey Questionnaire--2012 Hyattsville, MD: Division of Health Interview Statistics, National Center for Health Statistics; 2013 [July 3, 2014]. Available from: <a href="mailto:ftp://ftp.cdc.gov/pub/Health">ftp://ftp.cdc.gov/pub/Health</a> Statistics/NCHS/Survey Questionnaires/NHIS/2012/English.
- 26. Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB.
- 27. National Cancer Institute. Health Information National Trends Survey 4 (HINTS 4) Cycle 4 Questionnaire Bethesda, MD: National Cancer Institute; 2014 [cited 2016 November 1]. Available from: http://hints.cancer.gov/.
- 28. Colditz GA. Your Disease Risk. <a href="www.yourdiseaserisk.wustl.edu">www.yourdiseaserisk.wustl.edu</a> 2004 [cited 2015 September 17]. Available from: <a href="www.yourdiseaserisk.wustl.edu">www.yourdiseaserisk.wustl.edu</a>.
- 29. Colditz GA, Atwood KA, Emmons K, Monson RR, Willett WC, Trichopoulos D, Hunter DJ. Harvard report on cancer prevention volume 4: Harvard Cancer Risk Index. Risk Index Working Group, Harvard Center for Cancer Prevention. Cancer Causes Control. 2000;11(6):477-88. Epub 2000/07/06.

- 30. Rosner BA, Colditz GA, Hankinson SE, Sullivan-Halley J, Lacey JV, Jr., Bernstein L. Validation of Rosner-Colditz breast cancer incidence model using an independent data set, the California Teachers Study. Breast Cancer Res Treat. 2013;142(1):187-202. doi: 10.1007/s10549-013-2719-3. PMCID: PMC3825503.
- 31. Tait AR, Voepel-Lewis T, Zikmund-Fisher BJ, Fagerlin A. The effect of format on parents' understanding of the risks and benefits of clinical research: a comparison between text, tables, and graphics. Journal of health communication. 2010;15(5):487-501. doi: 10.1080/10810730.2010.492560. PMCID: PMC2915576.
- 32. National Cancer Institute. Health Information National Trends Survey 4 (HINTS 4) Cycle 3 Questionnaire Bethesda, MD: National Cancer Institute; 2014 [cited 2017 May 5]. Available from: http://hints.cancer.gov/.
- 33. National Cancer Institute. Health Information National Trends Survey 2005 Questionnaire Bethesda, MD: National Cancer Institute; 2005 [cited 2014 March 7]. Available from: http://hints.cancer.gov/.
- 34. Schwarzer R, Fuchs R. Self-efficacy and health behaviours. In: Conner M, Norman P, editors. Predicting Health Behaviour. Philadelphia, PA: Open University Press; 1995. p. 169-96.
- 35. National Cancer Institute. What does HINTS tell us about... Bethesda, MD: National Cancer Institute; 2014 [cited 2014 January 21]. Available from: <a href="http://hints.cancer.gov/topic.aspx">http://hints.cancer.gov/topic.aspx</a>.
- 36. Chung WW, Chen CA, Cupples LA, Roberts JS, Hiraki SC, Nair AK, Green RC, Stern RA. A New Scale Measuring Psychological Impact of Genetic Susceptibility Testing for Alzheimer's Disease. Alzheimer Dis Assoc Disord. 2009;23(1):50-6. PMCID: PMCPMC2743905.
- 37. Schwartz LM, Woloshin S, Black W, Welch G. The role of numeracy in understanding the benefit of screening mammography. Ann Intern Med. 1997;127(11):966-72.
- 38. Morris NS, MacLean CD, Chew LD, Littenberg B. The Single Item Literacy Screener: evaluation of a brief instrument to identify limited reading ability. BMC Fam Pract. 2006;7:21. doi: 10.1186/1471-2296-7-21. PMCID: PMC1435902.
- 39. Health NIfOSa. Quality of worklife questionnaire, 2010 2010 [cited 2017 May 5]. Available from: <a href="https://www.cdc.gov/niosh/topics/stress/pdfs/qwl2010.pdf">https://www.cdc.gov/niosh/topics/stress/pdfs/qwl2010.pdf</a>.
- 40. Weinstein ND, Atwood K, Puleo E, Fletcher R, Colditz G, Emmons KM. Colon cancer: Risk perceptions and risk communication. Journal of Health Communication. 2004;9:53-65.
- 41. Kotz D, Brown J, West R. Predictive validity of the Motivation To Stop Scale (MTSS): a single-item measure of motivation to stop smoking. Drug Alcohol Depend. 2013;128(1-2):15-9. doi: 10.1016/j.drugalcdep.2012.07.012.
- 42. McQueen A, Vernon SW, Swank PR. Construct Definition and Scale Development for Defensive Information Processing: An Application to Colorectal Cancer Screening. Health Psychol. 2013;32(2):190-202. Epub 2012/02/23. doi: 10.1037/a0027311.
- 43. Lukwago SN, Kreuter MW, Bucholtz DC, Holt CL, Clark EM. Development and validation of brief scales to measure collectivism, religiosity, racial pride, and time orientation in urban African American women. Fam Community Health. 2001;24(3):63-71.
- 44. Little TD, Schnabel KU, Baumert J. Modeling longitudinal and multilevel data: Practical issues, applied approaches, and specific examples. Mahwah, NJ: Psychology Press; 2000.
- 45. MacKinnon DP, Lockwood CM, Hoffman JM, West SG, Sheets V. A comparison of methods to test mediation and other intervening variable effects. Psychol Methods. 2002;7(1):83-104.
- 46. Rucker DD, Preacher KJ, Tormala ZL, Petty RE. Mediation analysis in social psychology: Current practices and new recommendations. Soc Personal Psychol Compass. 2011;5/6:359-71.
- 47. Bryan A, Schmiege SJ, Broaddus MR. Mediational analysis in HIV/AIDS research: estimating multivariate path analytic models in a structural equation modeling framework. AIDS Behavior. 2007;11(3):365-83.
- 48. Hayes AF, Scharkow M. The relative trustworthiness of inferential tests of the indirect effect in statistical mediation analysis: does method really matter? Psychol Sci. 2013;24(10):1918-27. doi: 10.1177/0956797613480187.
- 49. Hu L, Bentler PM. Evaluating model fit. In: Hoyle RH, editor. Structural Equation Modeling. Thousand Oaks, CA: Sage Publications; 1995. p. 76-99.
- 50. Hu L, Bentler PM. Cutoff criteria for fit indexes in covariance structure analysis: Conventional criteria versus new alternatives. Structural Equation Modeling. 1995(5):1-55.
- 51. Faul F. GPOWER Version 3.1.0. Kiel, Germany: Universitat Kiel; 2008. p. Software.
- 52. Faul F, Erdfelder E, Lang A-G, Buchner A. G\*Power 3: A flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007;39:175-91.

# **Special Considerations**

Not applicable.

# **List of Appendices**

Appendix A, Aim 2, Risk App Screens

Appendix C, Aim 2, Baseline Survey

Appendix D, Aim 2 Mental Imagery Script- Physical Activity

Appendix E, Aim 2 Mental Imagery Script- Sleep Hygiene Appendix F, Aim 2 Pamphlet

Appendix H, Aim 2 Intervention Screener

Appendix I, Aim 2 Participant Contact Sheet

Appendix J, Aim 2 Reminder Call Script

Appendix K, Aim 2 Screening Log

Appendix L, Aim 2 Baseline Survey 2 Physical Activity

Appendix M, Aim 2 Baseline Survey 2 Sleep Hygiene

Appendix N, Aim 2 Recruitment Call Script

Appendix O, Recruitment Email Script

Appendix P, Aim 2, BJC Ad

Appendix Q, Aim 2, Centerwatch Ad Appendix R, Aim 2, Facebook Posting

Appendix T, Aim 2, Website Posting

Appendix U, Aim 2, Reaserchmatch.org email

Appendix W, Aim 2 Data Collection Session 1 Guide

Appendix X Aim 2 Text Messages- Exercise

Appendix Y Aim 2 Text Messages- Sleep

Appendix Z, Aim 2 Final Survey Reminder Call Script

Appendix AA, Aim 2 Mailed Survey Invitation

Appendix BB, Aim 2 Final Follow-Up Survey

Appendix CC, Aim 2 Newspaper Advertisement

Appendix DD, Aim 2 Request Letter for SSN

Appendix EE, Aim 2 Gift card receipt

Appendix FF, Aim 2 Flyer

Appendix GG, Aim 2 Flyer Pull Tab

Appendix HH, Aim 2 Instructions for baseline survey

Appendix II, Aim 2 One year Follow Up Call Script with Questions

Appendix JJ, Aim 2 IRB Study Security Review 20170503-01

Appendix KK, Aim 2 Aws Security Whitepaper
Appendix LL, Aim 2 Twilio Whitepaper Security-Architecture